CLINICAL TRIAL: NCT03370328
Title: Essential Oils to Reduce Post-Operative Nausea and Vomiting
Brief Title: Reducing Up-set Stomach and Vomiting After Surgery Using Essential Oils
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Maxine Fearrington, Staff Nurse, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RSBR00069976
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Nausea
MeSH Terms: conditions — Nausea | interventions — peppermint oil; ginger extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peppermint oil (Experimental): post-op surgical patients
  Interventions: Other: Peppermint oil
- Ginger oil (Experimental): post-op surgical patients
  Interventions: Other: Ginger oil
- Peppermint and ginger oil (Experimental): post-op surgical patients
  Interventions: Other: Peppermint oil; Other: Ginger oil

INTERVENTIONS:
Other: Peppermint oil — The study product is a commercial essential oil product and nasal inhaler. It is to be prepared by a trained, independent individual who will add 4 drops of one of the three oils/oil combinations. The subject will be instructed to twist off the cap and position inhaler in such a way as to allow the subject to inhale the vapors; it can be reused for multiple administrations. Essential oils have been the subject of other studies in treating nausea. If nausea is unrelieved, treatment will progress to the ordered antiemetic.
  Arms: Peppermint and ginger oil; Peppermint oil
Other: Ginger oil — The study product is a commercial essential oil product and nasal inhaler. It is to be prepared by a trained, independent individual who will add 4 drops of one of the three oils/oil combinations. The subject will be instructed to twist off the cap and position inhaler in such a way as to allow the subject to inhale the vapors; it can be reused for multiple administrations. Essential oils have been the subject of other studies in treating nausea. If nausea is unrelieved, treatment will progress to the ordered antiemetic.
  Arms: Ginger oil; Peppermint and ginger oil

SUMMARY:
The purpose of this study is to determine if aromatherapy (essential oil) is effective at reducing up-set stomach and vomiting after surgery and in reducing the need for up-set stomach medications

DETAILED DESCRIPTION:
If participants decide to take part in this study, they will be asked to use choose a small nasal inhaler from a bag, open the sealed package, and inhale from the nasal inhaler 3 times, inhaling through the nose and exhaling through the mouth, just prior to entering the operating room. During recovery in the Post-operative acute care unit (PACU), nausea severity will be rated using a 0-3 scale where zero indicates no nausea.

If your score is 1-3, participants will be instructed/assisted in using a nasal inhaler 3 times, inhaling through the nose and exhaling through the mouth. After 5 minutes, nausea scores will be collected again and if the score is the same or higher, participants will be asked to use the nasal inhaler again in the same manner as before. If their nausea has not resolved after the second use, they will be give anti-nausea medication that a surgeon ordered. This process will be repeated again whenever you complain of nausea, until they are discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* post-op surgical patients at least 18 years of age or older
* the ability to understand and follow directions for use of essential oils
* the ability to understand and give informed consent to study
* the ability to understand, read and write English
* ambulatory or short-stay/23-hour patients

Exclusion Criteria:

* History of any pulmonary disease, including but not limited to: asthma, COPD, OSA, chronic bronchitis, pulmonary and ear, nose, throat (ENT) surgery patients
* Allergy to any of the ingredients in the essential oils
* Sensitivity to strong odors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Mean change in nausea score | baseline to 24 hours
  Nausea will be score on a scale of 0-3 with zero indicated no nausea.

CONTACTS AND LOCATIONS:
Overall Officials: Maxine Fearrington, MS, Principal Investigator — University of Rochester, Strong Memorial Hospital
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No